CLINICAL TRIAL: NCT01569997
Title: Interest of Systematic Tracking of Dementia Cases in Nursing Homes: Analysing the Contribution of MultiDisciplinary Team Meeting (MDTM) in Alzheimer's Disease and Related Diseases
Brief Title: Impact of Systematic Tracking of Dementia Cases on the Rate of Hospitalization in Emergency Care Units
Acronym: IDEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0910701; 2009-A01062-55 (Other: ID-RCB)
Record Dates: First submitted 2011-07-04; First posted 2012-04-04 (Estimated); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Dementia in Nursing Home
Keywords: Dementia; emergency hospitalization; nursing home; multidisciplinary meeting; cognitive decline; disability; residents; facilities; long term care unit; health policy; general practitioner; prevention
MeSH Terms: conditions — Dementia; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Other): Intervention group: nursing homes whose residents benefit from MDTM to identify the cases of dementia and to propose an adequate care project
  Interventions: Other: MultiDisciplinary Team Meetings (MDTM)
- control group (No Intervention): Control group: nursing homes whose residents continue to benefit from usual care

INTERVENTIONS:
Other: MultiDisciplinary Team Meetings (MDTM) — The MDTM, between the memory experts and Nursing Home coordinating practitioners, could help the nursing home medical staff identify the cases of dementia and propose these residents an adequate healthcare project (supplementary investigations, therapeutic modifications, hospitalizations...)
  Arms: Intervention group

SUMMARY:
Introduction: Epidemiological data show that in France only half of patients with Alzheimer disease are currently diagnosed in the general population. The absence of early diagnosis of dementia reduces the opportunities of patients to receive optimal care. One of the consequences of undiagnosed dementia is inadequate use of emergency care units.

The main objective: The main aim of this study is to evaluate the impact of a systematic case-finding procedure of dementia cases in nursing homes through a MDTM on the rate of hospitalization in emergency care units.

Secondary objectives:

To assess the impact of systematic tracking of dementia cases on the:

* Quantity and quality of drug-prescription
* Appropriateness of hospitalizations
* Prevalence of neuropsychiatric symptoms
* Dependency
* Quality of life
* Burden of nursing staff working conditions
* Planning of specific therapeutic measures
* Overall health care costs

DETAILED DESCRIPTION:
This is a multicentre, cluster randomized study comparing two parallel groups:

* Intervention group: nursing homes whose residents benefit from MDTM to identify the cases of dementia and to propose an adequate care project
* Control group: nursing homes whose residents continue to benefit from usual care In each group, 1000 elderly subjects aged over 60 years without documented diagnosis of dementia will be included and monitored for a period of 18 months.

Information about the main and secondary aims will be collected monthly through online questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Residents of both sex, aged 60 years or over
* Residents living in a nursing home participating in the study
* Residents living in the nursing home for 30 days or more
* Residents without diagnosed and documented dementia, identified as follows:

  * residents not identified by the French Healthcare system as suffering from dementia (ALD 15)
  * residents not benefiting from a specific care program or a specialized follow-up for dementia
  * residents for whom there is no appropriate investigation for dementia diagnosis in medical records
  * residents not taking specific drugs for dementia (Cholinesterase inhibitors and/or Memantine)
* Residents and their GP having received information about the study
* Residents and their GP having expressed their agreement to participate in the study

Exclusion Criteria:

* Residents aged less than 60 years
* Residents not living in a nursing home participating in study
* Residents living in nursing home for less than 30 days
* Residents with diagnosed and documented dementia, identified as follows:

  * residents Identified by the French Healthcare system as suffering from dementia (ALD 15)
  * residents benefiting from specific care programme or specialized follow-up for dementia
  * residents for whom there is appropriate investigation for dementia diagnosis in medical records
  * residents taking specific drugs for dementia (Cholinesterase inhibitors and/or Memantine)
* Residents and/or their GP who received no information about the study
* Residents and/or their GP having expressed their opposition to participate in the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1428 (Actual)
Dates: Start 2010-05; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Incidence of hospitalizations in emergency care units | 18 months
  Monthly collection during follow-up (18 months)

SECONDARY OUTCOMES:
Prevalence of antipsychotic prescription | Baseline visit, 4 months, 18 months
Incidence of inappropriate hospitalizations | 18 months
  Monthly collection during follow-up (18 months)
Prevalence of neuropsychiatric symptoms evaluated by NPI-nursing staff version | Baseline visit, 18 months
Dependency evaluated by AGGIR and IADL-4 items | Baseline visit, 18 months
Quality of life evaluated by QOL-AD | Baseline visit, 18 months
Number of nursing staff's time off work | 18 months
  Monthly collection during follow-up (18 months)
Number of days off work by nursing staff | 18 months
  Monthly collection during follow-up (18 months)
Presence of advanced care planning in patients medical records | Baseline visit, 18 months
  Advanced care planning will be checked through behavioural disosders, transfer to hospital intensive care and resuscitation
Overall healthcare costs | 18 months
  Monthly collection during follow-up (18 months)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre ALLAN, MD, Principal Investigator — EHPAD MAISON DE RETRAITE SAINT JOSEPH - MAZAMET; Véronique ARNAUD-ULLIET, MD, Principal Investigator — EHPAD MA MAISON MONTPELLIER
Locations (90):
- France (90):
  - Centre de Gerontologie Pompeyrie Chu Agen, Agen
  - Ehpad Maison de Retraite Louise Anceau, Albi
  - Ehpad Maison de Retraite Olga Ducoudray, Albi
  - Ehpad Mr "Les Jardins de Jouvence", Albi
  - Mapad La Renaudie Ch Albi, Albi
  - Ehpad Les Ajoncs D'Or, Allaire
  - Ehpad Maison de Retraite Hl Ax Les Thermes, Ax-les-Thermes
  - Ehpad Marie Lehman, Balma
  - Ehpad Kerdigemer, Brest
  - Ehpad Residence Ker-Heol, Brest
  - Ehpad Residence Saint Astier, Catus
  - Mapa de L'Hopital Local de Caussade, Caussade
  - Ehpad Maison de Retraite Ste Marthe, Ceignac
  - EHPAD Résidence Castelgirou, Cépet
  - Ehpad Leon Ronzier Joly, Clermont-l'Hérault
  - Ehpad Themis Lasplanes, Colomiers
  - Ehpad Maison de Retraite Joseph Sauvy, Err
  - Ehpad Residence Borde Haute Promo-Accueil, Escalquens
  - Mapad "Firmi", Firmi
  - Ehpad Hopital Local Fleurance, Fleurance
  - Ehpad Mr Bellissen Chi Du Val D'Ariege, Foix
  - Ehpad Dr Robert, Guer
  - Ehpad Residence Grand'Maison, L'Union
  - Ehpad Residence Provencale Medicafrance, La Roquebrussanne
  - Ehpad Residence Clairefontaine, Lamorlaye
  - Mapad Ch Lavaur, Lavaur
  - Ehpad Saint Reah Hir, Le Conquet
  - Ehpad Residence D'Automne de La Ferme, Le Mée-sur-Seine
  - Ehpad Maison de Retraite "Les Charmilles", Lescure-d'Albigeois
  - Residence Le Parc, Lézat-sur-Lèze
  - Ehpad La Cheneraie, Lherm
  - Ehpad Mr Lagrange, Lisle-sur-Tarn
  - Mapad Labastide Ch Lourdes, Lourdes
  - Ehpad Emile Dubois, Marchiennes
  - Ehpad Les Mille Soleils, Marciac
  - Ehpad Et. Public Gerontologie de Marines, Marines
  - AP-HM Hôptal La Timone Service de Pédiatrie Mutidisciplinaire, Marseille
  - Ehpad Maison Retraite Hl Mauvezin, Mauvezin
  - Ehpad Maison de Retraite Saint Joseph, Mazamet
  - Ehpad Maison de Retraite Privee de Mazeres, Mazères
  - Ehpad L'Ecrin Des Sages, Mèze
  - Ehpad-Maison Retraite Hl Mirande, Mirande
  - Ehpad Chis Castelsarrasin-Moissac, Moissac
  - Ehpad Maison Retraite Ch Montauban, Montauban
  - Ehpad Era Caso, Montauban-de-Luchon
  - Ehpad Ma Maison, Montpellier
  - Ehpad Maison de Retraite Sainte Agnes, Montredon-Labessonnié
  - Ehpad L'Acacia, Nailloux
  - Logements Foyer La Fontanelle, Naucelle
  - Ehpad Fondation Pauliani, Nice
  - Ehpad Les Noisetiers, Nice
  - Ehpad Residence Ancilla, Nice
  - Ehpad Mais de Retraite Saint-Joseph, Ossun
  - Ehpad Mr Bariol Chi Du Val D'Ariege, Pamiers
  - Ehpad Residence Le Parc, Panazol
  - AP-HP Hôpital Necker Enfants Malades Service d'endocrinologie pédiatrique - 149 route de Sèvres, Paris
  - Ehpad Furtado Heine, Paris
  - Ehpad Julie Siegfried, Paris
  - Ehpad La Pirandelle, Paris
  - Ehpad Residence Anselme, Paris
  - Ehpad Residence Belleville, Paris
  - Ehpad Residence Herold, Paris
  - Ehpad Residence Oceane, Paris
  - Ehpad Tiers Temps Paris, Paris
  - Ehpad Residence Adeline, Pierre-Buffière
  - Ehpad Residence D'Automne Medica-France, Reims
  - Ehpad L'Oree Du Bois, Rieux-Volvestre
  - Ehpad Residence Saint-Amans, Rodez
  - Ehpad Le Jardin Des Loges, Saint-Bonnet
  - Ehpad Maison Retraite Orelia Ch St Gaudens, Saint-Gaudens
  - Ehpad Residence Themis La Joie de Vivre, Saint-Lys
  - Ehpad Genevriers, Saint-Martory
  - Ehpad A Labouilhe, Saint-Orens-de-Gameville
  - Ehpad Public de Saint-Remy de Provence, Saint-Rémy-de-Provence
  - Ehpad Les Bruyeres, Sousceyrac
  - Ehpad Maison de Retraite Chic Tarbes Vic, Tarbes
  - Ehpad Residence "Le Doyenne Du Carmel", Tarbes
  - Ehpad Sainte Anne, Tinténiac
  - Ehpad de La Cote Pavee, Toulouse
  - Ehpad Gaubert, Toulouse
  - Ehpad Mr Henri Iv, Toulouse
  - Ehpad Pierre Ducis, Toulouse
  - Ehpad Residence La Cotonniere, Toulouse
  - Ehpad Residence Le Clos Des Carmes, Toulouse
  - Ehpad Residence Marguerite, Toulouse
  - Ehpad Residence Saint-Simon, Toulouse
  - Usld Domaine de La Cadene, Toulouse
  - Ehpad Umt, Valence-d'Albigeois
  - Ehpad Maisonneuve, Villefranche-de-Lauragais
  - Ehpad Saint-Jacques, Villemur-sur-Tarn

REFERENCES:
- [Result] Rolland Y, Tavassoli N, de Souto Barreto P, Perrin A, Laffon de Mazieres C, Rapp T, Hermabessiere S, Tournay E, Vellas B, Andrieu S. Systematic Dementia Screening by Multidisciplinary Team Meetings in Nursing Homes for Reducing Emergency Department Transfers: The IDEM Cluster Randomized Clinical Trial. JAMA Netw Open. 2020 Feb 5;3(2):e200049. doi: 10.1001/jamanetworkopen.2020.0049. PMID 32101308